CLINICAL TRIAL: NCT02979834
Title: A Frequently Asked Question: When Will I Feel The First Movements of My Baby?
Brief Title: When Will I Feel The First Movements of My Baby?
Acronym: FFM
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hatice Akkaya, Principle investigator, Kayseri Education and Research Hospital
Other Study IDs: E52332816/53
Record Dates: First submitted 2016-11-26; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Early Pregnancy
Keywords: fetal movement; placenta site; body mass index; maternal education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Early perception group: The group with early perception of fetal movement (<25th percentile)
- Average perception group: The group with average perception of fetal movement (>25th and <75th percentile)
- Late perception group: The group which late perception of fetal movement (>75 percentile)

SUMMARY:
This study aims to investigate average gestational week in which mothers feel the babies'movements for the first time and maternal-fetal factors affecting this time.

DETAILED DESCRIPTION:
Most of the obstetricians face the question; "When Will I Feel The First Movements of My Baby?", in daily practice. It becomes a challenge for the obstetrician to answer this question. Because, there is not a sufficient data in the current literature on this issue. A broad range of weeks for fetal quickening are reported as 16th to 20th weeks, in round figures. So, when a woman in the 21st gestational week , asks this question to the obstetrician and informed according to aforementioned literature knowledge, the woman will ask another question immediately after: "What is the problem with my baby?". But, the obstetrician will not be able to give an assuring answer because of the lack of knowledge in the current literature.Thus, to cope with such a clinical situation, the investigators decided to investigate the average week in which pregnant women in a low risk population, felt the babies' movements for the first time and to find out the affects of probable factors which may act on this time.

ELIGIBILITY:
Inclusion Criteria:

* The study population included spontaneous, singleton pregnancies at first and second-trimester of their pregnancy

Exclusion Criteria:

* Multiple pregnancies, evidence of fetal or maternal infection, hypertensive disorders of gestation, gestational and pregestational diabetes mellitus, maternal drug use, evidence of fetal congenital abnormalities and amniotic fluid abnormalities were stated as the exclusion criteria for the study group.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three groups were formed according to the gestational week in which fetal movements felt by mother for the first time. 25th percentile, 50thand 75th percentile values were determined .Participants who felt the babies' movements at or before 25th percentile value constituted Group1 or early perception group, participants who felt the babies' movements between 25th and 75th percentile value constituted Group 2 or average perception group and the participants who felt the babies'movements at or beyond 75th value constituted Group 3 or late perception group. Subsequently, these three groups were compared regarding maternal age, gestational week of inclusion in the study, obstetric features, maternal body mass index values, caffeine consumption, smoking status, maternal education status, placental localization and fetal gender.
Sampling Method: Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
placental settlement via ultrasound | 5 minutes
  Relationship between placental location obtained via sonography and fetal movement perception

SECONDARY OUTCOMES:
maternal body mass index measurement | 3 minutes
  Relationship between Maternal Body Mass Index calculated by dividing body weight to height and fetal movement perception
maternal age | 1 minute
  Relationship between Maternal age according to questionnaire and fetal movement perception
parity | 1 minute
  Relationship between Maternal parity according to questionnaire and fetal movement perception
educational status | 1 minute
  Relationship between maternal education status according to questionnaire and fetal movement perception
smoking | 1 minute
  Relationship between Maternal smoking according to questionnaire and fetal movement perception
tea and coffee consumption | 1 minute
  Relationship between maternal tea and coffee conception according to questionnaire and fetal movement perception
fetal gender | 5 minutes
  Relationship between fetal gender obtained via sonography and fetal movement perception
regular pregnancy follow ups | 1 minute
  Relationship between regular pregnancy follow ups recorded on patient record system and fetal movement perception

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Akkaya, M.D, Principal Investigator — Kayseri Education and Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
The data belonging to participant will be available to any researcher or editorial review board if needed.